CLINICAL TRIAL: NCT06878599
Title: Intratympanic Injection of Dexamethasone With Hyaluronic Acid in Treatment of Sudden Sensorineural Hearing Loss
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Essam Ali AbuElmagd, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hyaluronic acid in SSNHL
Record Dates: First submitted 2025-03-08; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sudden Sensorineural Hearing Loss (SSNHL)
Keywords: Hyaluronic acid; Dexamethasone; SSNHL; Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Hyaluronic Acid; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyalouronic acid with dexamethasone injection (Experimental): Intratympanic injection
  Interventions: Combination Product: Hyaluronic Acid (HA); Drug: Dexamethasone
- Dexamethasone injection (Active Comparator): Intratympanic injection
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Combination Product: Hyaluronic Acid (HA) — Adding Hyaluronic acid to dexamethasone as intratympanic injection
  Arms: Hyalouronic acid with dexamethasone injection
Drug: Dexamethasone — Intratympanic injection of Dexamethasone

SUMMARY:
* To evaluate efficacy of intratympanic injection of dexamethasone and hyaluronic acid mixture as a treatment modality in cases of sudden sensorineural hearing loss (SSNHL).
* To compare outcomes of intratympanic injection of dexamethasone and hyaluronic acid mixture to dexamethasone alone in treatment of SSNHL.

DETAILED DESCRIPTION:
Sudden sensory neural hearing loss (SSNHL) is defined as sensorineural hearing loss of at least 30 dB over 3 consecutive frequencies within 3 days. Different treatment modalities have been used in treatment of SSNHL including systemic corticosteroids alone or in combination with vasodilators as pentoxifylline and hydroxyethylstarch (HES) or low molecular weight dextran, hyperbaric oxygen therapy & plasmapheresis.

Intratympanic (IT) dexamethasone application has shown significantly higher perilymph steroid concentrations with lower systemic concentrations, thus avoiding the side effects associated with the systemic route. It has been used with varying results for the treatment of Meniere's disease, SSNHL, low frequency hearing loss and tinnitus. After IT injection, the drug concentration in the inner ear depends on the drug being in contact with the round window membrane (RWM), absorbing it from the middle ear into the inner ear. However, large amount of the injected drugs are either absorbed by the middle ear mucosa or evacuated via the eustachian tube.

It has been postulated that combining the drug with a biodegradable material will prolong its availability in the middle ear and/or aid its diffusion across the RWM. Between these materials, Hyaluronic acid (HA) is a natural product normally present is humans' perilymph in small amounts along with many other tissues throughout the body. Several postulations have been given to HA mechanism of action in drug delivery in the middle ear either by its osmotic effect on the perilymph, modulating RWM permeability or altering blood viscosity thus increasing blood and oxygen delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 18 and over)
2. Patients with sudden sensory neural hearing loss (SSNHL)

Exclusion Criteria:

1. Patients with middle or external ear pathology.
2. Patient with history of traumatic skull base fracture.
3. Patients with previous ear surgery.
4. Patients with other neurological symptoms or signs (Other cranial nerves affection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Degree of hearing improvement | From the start of injections to 4 weeks after the end of injections
  Using Pure Tone Audiometry (PTA), patients will be assessed once prior to the start of intratympanic injections, at its end and 4 weeks after. A 30 dB improvement in bone conduction threshold (BCT) in PTA is considered a significant improvement, while improvements of 10-30 dB and >10 dB are considered as partial recovery and non-recovery respectively.
Assessing each frequency difference | From the start of injections to 4 weeks after the end of injections
  Assessment will also measure the differences in each frequency independently between the pre and post treatment PTA.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt